CLINICAL TRIAL: NCT04485390
Title: Impact of the Organization of the First Responders in the Remote Areas on Cardiac Arrest Victim Survival: an Utstein Analysis
Brief Title: Impact of the Organization of the First Responders in the Remote Areas on Cardiac Arrest Victim Survival
Status: Completed | Type: Observational
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Matej Strnad, Assoc. Professor, University Medical Centre Maribor
Other Study IDs: UKC-MB-KME-24/20
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Cardiac Arrest, Sudden
Keywords: cardiac arrest; cardiopulmonary resuscitation; automated external defibrillator; first responders
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First responder group: Cardiac arrest victims in remote areas resuscitated by the first responders before the arrival of the EMS.
  Interventions: Other: Basic life support witn use of an AED before EMS
- EMS groups: Cardiac arrest victims in remote areas resuscitated by the EMS.

INTERVENTIONS:
Other: Basic life support witn use of an AED before EMS — BLS performance with use of an AED before arrival of EMS
  Groups: First responder group

SUMMARY:
Emergency medical services (EMS) provide emergency care not only in the urban but also in the remote areas which could be up to 40 minutes from the EMS station. Thus, a cardiac arrest victim in those remote areas has a low likelihood to survive the cardiopulmonary resuscitation. Therefore, we have organized first responders (who are mostly volunteer fire-fighters) in the remote areas and taught them how to perform basic life support (BLS) with use of an automated external defibrillator (AED). In the case of a cardiac arrest the medical dispatcher activates simultaneously the EMS and the first responders, who perform the BLS with the use of an AED before the arrival of EMS.

The aim of the study is to analyze and compare the survival of the cardiac arrest victims in remote areas in the time period when the first responders were not organized yet compared to the time period when the first responders were activated to perform BLS.

ELIGIBILITY:
Inclusion Criteria:

* cardiac arrest in adult victims

Exclusion Criteria:

* cardiac arrest in pediatric population

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In the study will be included all adult cardiac arrest victims in the remote areas.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Return of spontaneous circulation (ROSC) | 5 years
  The number of patients who gained the ROSC.
Survival to hospital discharge | 5 years
  The number of patients who survived to hospital discharge.
Neurological outcome | 5 years
  The number of patients with good neurological outcome assessed with cerebral performance score (CPC 1-2).

SECONDARY OUTCOMES:
Survival till hospital admission | 5 years
  The number of patients who survived to hospital admission.
30 day survival | 5 years
  The number of patients who survived first 30 days after cardiac arrest.

IPD SHARING:
Plan to Share IPD: Undecided